CLINICAL TRIAL: NCT05467670
Title: Safety and Efficacy of Anti-CD47, ALX148 in Combination with Liposomal Doxorubicin and Pembrolizumab in Patients with Recurrent Platinum-resistant Ovarian Cancer: Phase II Study
Brief Title: Safety and Efficacy of Anti-CD47, ALX148 in Combination with Liposomal Doxorubicin and Pembrolizumab in Recurrent Platinum-resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander B Olawaiye, MD (Other)
Collaborators: ALX Oncology (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Alexander B Olawaiye, MD, Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-193
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: anti-CD47 therapy; platinum resistance; macrophage mediated phagocytosis; checkpoint inhibitors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; ALX148; Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALX148 + Doxorubicin (PLD) + Pembrolizumab (Experimental): Given on Day 1 of each 21 day cycle, in the following order of administration:
  200 mg IV pembrolizumab* (maximum of 2 years (approximately 35 cycles)
  45 mg/kg IV ALX148
  30 mg/m^2 IV doxorubicin (Pegylated Liposomal Doxorubicin (PLD)*
  *standard of care
  Interventions: Drug: Pembrolizumab; Drug: ALX148; Drug: Doxorubicin

INTERVENTIONS:
Drug: Pembrolizumab — A type of immunotherapy that stimulates the body's immune system to fight cancer cells by targeting and blocking PD-1 proteins on the surface of certain immune T-cells, thus triggering the T-cells to find and kill cancer cells.
  Other Names: Keytruda®
Drug: ALX148 — A fusion protein comprised of a high affinity CD47 blocker linked to an inactive immunoglobulin Fc region, enhancing innate and adaptive immune responses against cancer.
  Other Names: evorpacept
Drug: Doxorubicin — An anthracycline that slows/stops the growth of cancer cells by blocking an enzyme called topo isomerase 2, used as second line non-platinum chemotherapy in patients with platinum-resistant ovarian cancer.
  Other Names: (Pegylated Liposomal Doxorubicin (PLD)

SUMMARY:
Immunotherapy with immune checkpoint inhibitors, including pembrolizumab, have emerged as a promising option in several solid cancers with durable effect and low toxicity profile. However, the benefit is limited to smaller subset of solid tumors. This trial involves the enhancement of current immune checkpoint-based immunotherapy with ALX148, an agent that inhibits CD47 (a trans-membrane protein that is highly expressed on the surface of many solid tumors as compared to normal cells).

DETAILED DESCRIPTION:
All patients on this study will receive Pegylated Liposomal Doxorubicin (PLD) as standard of care combined with pembrolizumab and ALX148 iv every 21 days. Treatment of 45 mg/kg Q3W ALX148 in combination with pembrolizumab + chemotherapy will continue until disease progression or unacceptable grade 3/4 toxicities. For patients with a complete response to therapy, maintenance therapy with pembrolizumab and ALX148 will be continued for 12 months. Patients will have up to 4 weeks of screening, and will be treated until disease progression, patient withdraws consent, unacceptable toxicity occurs, complete response or the study is terminated. Patients may continue treatment after radiographic progression if, in the judgment of the treating investigator the patient is deriving clinical benefit from study treatment by demonstrating an absence of clinical symptoms or signs indicating clinically significant disease progression; no decline in performance status; absence of rapid disease progression or threat to vital organs or critical anatomical sites. A follow-up visit will occur within between 28 days and 35 days after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have recurrent epithelial ovarian cancer.
2. Platinum-resistant disease: Patients who recur within < 6 months of prior platinum-based therapy excluding those with primary platinum refractory disease (see exclusion criteria).
3. Following histology types are acceptable: high grade serous or high grade endometrioid, clear cells, high grade translational cell, poorly differentiated or undifferentiated carcinomas, mixed histology (including one of above histology).
4. 0-3 prior lines in platinum-resistant setting.
5. Known BRCA status or willing to be tested.
6. Up to 5 prior lines of therapy are allowed.
7. Participants must have measurable disease based on RECIST 1.1 with at least one target lesion.
8. Participants must have an ECOG performance status of 0-1.
9. Participants must be female, Age >18 years. Because no dosing or AE data are currently available on the use of pembrolizumab in combination with ALX148 in participants ≤18 years of age, children are excluded from this study.
10. Participants must have normal organ and marrow function as defined below within 14 days of enrollment unless otherwise indicated.
11. Participants must have the ability to understand and the willingness to sign a written informed consent document.
12. Negative serum or urine pregnancy test at screening for women of childbearing potential.
13. Willing to use highly effective contraception throughout the study and for at least 4 months after last treatment administration if childbearing potential exists.
14. Availability of an archival FFPE tumor tissue block from primary diagnosis specimen, metastatic, or recurrent site. If an FFPE tissue block cannot be provided then 15 unstained slides (10 microns, 10 slides minimum) will be acceptable. Please refer to the laboratory manual for complete details.

Exclusion Criteria:

1. Patients with sarcoma or carcinosarcoma or low-grade carcinoma.
2. Patients with primary platinum-refractory carcinoma who progressed while on or within 3 months of primary platinum-based combination therapy at first line setting.
3. Prior systemic anti-cancer therapy including investigational agents within 4 weeks [can be in follow-up phase of prior study and could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to [randomization /allocation]. AEs due to previous therapies will be evaluated for eligibility. Recovery from complications due to prior must be adequate.
4. Prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
6. Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable with no evidence of disease progression for 3 months.
7. Patients having received prior therapy with PD1, PDL1, CTLA4 inhibitors, CD47 or SIRP1- α inhibitors or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137), or other immunotherapeutic agents.
8. Prior therapy with PLD. Patients who received PLD in combination with platinum in platinum sensitive setting are allowed if they had initial objective complete response and PLD-platinum free interval of 6 months or more.
9. Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing ≥ 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Patients currently on immunosuppressive therapy except: intra-nasal, inhaled, topical or local steroid injections, steroids as premedication, systemic corticosteroids ≤10 mg/day of prednisone or equivalent
13. Patients who are pregnant or breast feeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
14. Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis ((non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease), pulmonary fibrosis.
15. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
16. Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and underwent potentially curative therapy: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. Patients with a history of carcinoma in situ of the bladder are excluded.
17. Prior organ transplantation including allogenic stem-cell transplantation.
18. Active infection requiring intravenous systemic therapy. Oral antibiotic therapy is allowed.
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

    Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority or treating physician per standard of care except patients with a known history of Hepatitis B not on a stable dose of antiviral therapy, with HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
20. History of infection with (screening tests not required) human immunodeficiency virus; except following situation:

    a. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible for this trial.
21. Received live or live-attenuated vaccine within 4 weeks of the first dose of treatment and while on trials is prohibited except for administration of inactivated vaccines. Influzena and COVID vaccinations are permissible.
22. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade ≥ 3).
23. Persistent toxicity related to prior therapy (NCI CTCAE v. 5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
24. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
25. A WOCBP who has a positive urine pregnancy test within 72 hours prior to [randomization/allocation] (see Appendix IV). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years (cohort)
  The proportion of patients having either a complete response (CR) or partial response (PR), per RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. For non-target lesions, CR is the disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  The number of months from the date of study enrollment until date of death ( from any cause) or last known date of follow up if otherwise lost to follow up.
Progression-free survival (PFS) | Up to 5 years
  The number of months from the date of study enrollment to the date of an event of disease progression (per RECIST 1.1) or to the date of death from any cause. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Objective response rate Immune-related Response Criteria (iRECIST) | Up to 3 years (cohort)
  The proportion of patients with complete or partial response per iRECIST. irCR (Complete Response):Disappearance of non-nodal lesions. All pathologic lymph nodes <10 mm (2 consecutive measures ≥4 weeks apart); irPR (Partial Response):≥30% decrease from baseline (2 consecutive measures ≥4 weeks apart); All pathologic lymph nodes <10 mm (Non-Target Lesions: Any other than disappearance of all non-nodal lesions and reduction of pathologic lymph nodes <10 mm). Baseline tumor burden: sum of single diameters (short axis for nodal lesions, longest diameter for other lesions) for target lesions. In subsequent scans, the diameters of new measurable lesions are added to the tumor burden. Re-treatment: ≤5 target lesions (=/≠ original lesions) are selected and a new baseline tumor burden will be established.
Duration of response (DOR) | Up to 3 years (cohort); at 12 weeks (patient)
  The number of months from the date of study enrollment to the date of disease progression or death in those participants who achieve complete or partial response per RECISIT 1.1. Complete Response (CR): Disappearance of all target lesions. For non-target lesions, CR is the disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change not a single lesion increase.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander B Olawaiye, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No